CLINICAL TRIAL: NCT02691507
Title: A Clinical Trial to Determine the Therapeutic Benefit of an Investigational Over-The-Counter Cream on Dry, Itchy Skin of Adults and Children With Atopic Dermatitis.
Brief Title: Trial to Determine the Therapeutic Benefit of an OTC Cream on Dry, Itchy Skin of Adults and Children With Eczema
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johnson & Johnson Consumer Inc. (J&JCI) (Industry)
Responsible Party: Sponsor
Organization: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CO - 151102105611 - SACT
Record Dates: First submitted 2016-02-22; First posted 2016-02-25 (Estimated); Results first posted 2017-03-06 (Actual); Last update posted 2017-03-06 (Actual); Status verified 2017-01

CONDITIONS: Atopic Dermatitis
Keywords: Eczema, Itchy Skin
MeSH Terms: conditions — Dermatitis, Atopic; Eczema; Pruritus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Positive Control (Active Comparator): Marketed - EpiCeram(R) Skin Barrier Emulsion: Apply in a thin layer to the affected skin areas 2 times per day (or as needed) and massage gently into the skin.
  Interventions: Device: EpiCeram Skin Barrier Emulsion
- Experimental (Experimental): Not Yet Marketed - 1% Colloidal Oatmeal Balm: Apply at least once per night or more if needed.
  Interventions: Drug: Experimental Product 1% Colloidal Oatmeal Balm

INTERVENTIONS:
Device: EpiCeram Skin Barrier Emulsion — EpiCeram Skin Barrier Emulsion
  Arms: Positive Control
Drug: Experimental Product 1% Colloidal Oatmeal Balm — Experimental Product 1% Colloidal Oatmeal Balm
  Other Names: Eczema Moisturizing Balm
  Arms: Experimental

SUMMARY:
The objective of this 1 week trial is to evaluate the efficacy of an over-the-counter (OTC) 1% colloidal oatmeal skin protectant cream in adults and children with mild to moderate AD.

DETAILED DESCRIPTION:
Approximately 60 subjects will be enrolled to ensure 52 subjects complete the study (39 subjects: active treatment and 13 subjects: positive control).

Adults and children (ages 12 and over) will receive either a marketed or not yet marketed investigational product for the treatment of eczema. Subjects will be asked to stop use of prescription and all eczema treatments 2 days before the start of the study and during the study. Subjects will apply study product as indicated for 7 days to affected areas.

Subjects will record treatment use in a daily diary and complete questionnaires. A dermatologist will examine and score the eczema and symptoms. Skin moisture levels will also be tested.

ELIGIBILITY:
Inclusion Criteria:

1. Able to comprehend and follow the requirements of the study (including availability on scheduled visit dates)
2. Male or female of any race or ethnicity, ages 12 and older
3. Diagnosed as having eczema
4. Willing to stop use of all non-assigned moisturizers and/or creams for the entire duration of the study

Exclusion Criteria:

1. Known sensitivity to any investigational product ingredient
2. Females who are pregnant , breastfeeding , or planning on becoming pregnant during the study
3. Individuals with a history of skin cancer
4. Use of a therapeutic (over-the-counter or prescription) body wash that contains an active ingredient for eczema
5. Participation in any clinical study within 30 days of Visit 1
6. Active infection of any type at the start of the study
7. Diagnosed as having severe eczema
8. Has a compromised immune system
9. Individuals with any planned surgeries and/or invasive medical procedures during the course of the study
10. Requires greater than 2.0mg/day inhaled or intranasal corticosteroids

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2016-02; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amisha Parikh-Das, PhD, Study Director — Johnson & Johnson Consumer Inc. (J&JCI); Lily Jiang, PhD, Principal Investigator — Stephens & Associates, Inc (Texas Research Center); Kun M Qian, MD, Principal Investigator — Stephens & Associates, Inc (Colorado Research Center)
Locations (2):
- United States (2):
  - Stephens & Associates (Colorado Research Center), Colorado Springs, Colorado
  - Stephens & Associates (Texas Reserach Center), Richardson, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- 1% Colloidal Oatmeal Balm: 1% colloidal oatmeal balm applied in a thin layer to affected skin areas at least once per day (or as needed)
- EpiCeram Skin Barrier Emulsion: EpiCeram skin barrier emulsion applied in a thin layer to affected skin areas two times per day (or as needed)
Period: Overall Study
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Started | 40 | 13
Completed | 40 | 12
Not Completed | 0 | 1
Not completed — Missed Visit 3 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion | Total
Number analyzed (Participants) | 40 | 13 | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.0 (17.43) | 45.5 (18.51) | 43.6 (17.55)
Gender [Count of Participants; unit: Participants]
  Female | 25 | 9 | 34
  Male | 15 | 4 | 19
Region of Enrollment [Number; unit: participants]
  United States | 40 | 13 | 53

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Itch Assessment Score Immediately Following Treatment
Description: The severity of the itch was assessed by the subject using a 0-10 cm visual analog scale (VAS) where 0 = no itch and 10 = worst itch imaginable.
Time Frame: Baseline to immediately following treatment
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 40 | 13
units on a scale | 1.93 (2.753) | 2.64 (2.482)
Statistical Analysis 1: Comparison: 1% Colloidal Oatmeal Balm; The null hypothesis was no difference between the baseline score and the post-baseline score. The alternative hypothesis was a difference between the baseline score and the post-baseline score; Test type: Superiority or Other; p < 0.001, Paired t-test — The significance level threshold level was 0.05
Statistical Analysis 2: Comparison: EpiCeram Skin Barrier Emulsion; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.002, Paired t-test — The significance level threshold level was 0.05
Statistical Analysis 3: Comparison: 1% Colloidal Oatmeal Balm vs EpiCeram Skin Barrier Emulsion; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.616, ANCOVA — The significance level threshold level was 0.05; Change from baseline as response, baseline score as covariate and treatment as factor; Mean Difference (Final Values) = 0.40, 95% CI 2-sided [-1.196 to 1.998], Standard Error of Mean 0.795

2. Primary Outcome: Change From Baseline in the Itch Assessment Score 1 Hour After Treatment
Description: as for outcome 1
Time Frame: Baseline to one hour after treatment
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 40 | 13
units on a scale | 3.00 (2.624) | 3.08 (2.559)
Statistical Analysis 1: Comparison: 1% Colloidal Oatmeal Balm; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Paired t-test — The significance level threshold level was 0.05
Statistical Analysis 2: Comparison: EpiCeram Skin Barrier Emulsion; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Paired t-test — The significance level threshold level was 0.05
Statistical Analysis 3: Comparison: 1% Colloidal Oatmeal Balm vs EpiCeram Skin Barrier Emulsion; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.297, ANCOVA — The significance level threshold level was 0.05; Change from baseline as response, baseline score as covariate and treatment as factor; Mean Difference (Final Values) = 0.85, 95% CI 2-sided [-0.767 to 2.460], Standard Error of Mean 0.803

3. Primary Outcome: Change From Baseline in the Itch Assessment Score 2 Hours After Treatment
Description: as for outcome 1
Time Frame: Baseline to two hours after treatment
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 40 | 13
units on a scale | 3.46 (2.849) | 3.65 (2.236)
Statistical Analysis 1: Comparison: 1% Colloidal Oatmeal Balm; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Paired t-test — The significance level threshold level was 0.05
Statistical Analysis 2: Comparison: EpiCeram Skin Barrier Emulsion; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Paired t-test — The significance level threshold level was 0.05
Statistical Analysis 3: Comparison: 1% Colloidal Oatmeal Balm vs EpiCeram Skin Barrier Emulsion; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.394, ANCOVA — The significance level threshold level was 0.05; Change from baseline as response, baseline score as covariate and treatment as factor; Mean Difference (Final Values) = 0.73, 95% CI 2-sided [-0.973 to 2.426], Standard Error of Mean 0.846

4. Primary Outcome: Change From Baseline in the Itch Assessment Score 3 Hours After Treatment
Description: as for outcome 1
Time Frame: Baseline to three hours after treatment
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 38 | 13
units on a scale | 3.93 (2.635) | 4.88 (2.094)
Statistical Analysis 1: Comparison: 1% Colloidal Oatmeal Balm; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Paired t-test — The significance level threshold level was 0.05
Statistical Analysis 2: Comparison: EpiCeram Skin Barrier Emulsion; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Paired t-test — The significance level threshold level was 0.05
Statistical Analysis 3: Comparison: 1% Colloidal Oatmeal Balm vs EpiCeram Skin Barrier Emulsion; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.690, ANCOVA — The significance level threshold level was 0.05; Change from baseline as response, baseline score as covariate and treatment as factor; Mean Difference (Final Values) = 0.28, 95% CI 2-sided [-1.140 to 1.709], Standard Error of Mean 0.708

5. Primary Outcome: Change From Baseline in the Itch Assessment Score 4 Hours After Treatment
Description: as for outcome 1
Time Frame: Baseline to four hours after treatment
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 40 | 13
units on a scale | 3.85 (2.580) | 4.92 (2.048)
Statistical Analysis 1: Comparison: 1% Colloidal Oatmeal Balm; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Paired t-test — The significance level threshold level was 0.05
Statistical Analysis 2: Comparison: EpiCeram Skin Barrier Emulsion; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Paired t-test — The significance level threshold level was 0.05
Statistical Analysis 3: Comparison: 1% Colloidal Oatmeal Balm vs EpiCeram Skin Barrier Emulsion; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.914, ANCOVA — The significance level threshold level was 0.05; Change from baseline as response, baseline score as covariate and treatment as factor; Mean Difference (Final Values) = -0.08, 95% CI 2-sided [-1.556 to 1.397], Standard Error of Mean 0.735

6. Primary Outcome: Change From Baseline in the Itch Assessment Score 5 Hours After Treatment
Description: as for outcome 1
Time Frame: Baseline to five hours after treatment
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 40 | 13
units on a scale | 4.06 (2.721) | 5.25 (1.846)
Statistical Analysis 1: Comparison: 1% Colloidal Oatmeal Balm; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Paired t-test — The significance level threshold level was 0.05
Statistical Analysis 2: Comparison: EpiCeram Skin Barrier Emulsion; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Paired t-test — The significance level threshold level was 0.05
Statistical Analysis 3: Comparison: 1% Colloidal Oatmeal Balm vs EpiCeram Skin Barrier Emulsion; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.757, ANCOVA — The significance level threshold level was 0.05; Change from baseline as response, baseline score as covariate and treatment as factor; Mean Difference (Final Values) = -0.24, 95% CI 2-sided [-1.796 to 1.314], Standard Error of Mean 0.774

7. Primary Outcome: Change From Baseline in the Itch Assessment Score 6 Hours After Treatment
Description: as for outcome 1
Time Frame: Baseline to six hours after treatment
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 40 | 13
units on a scale | 4.07 (2.824) | 5.55 (1.884)
Statistical Analysis 1: Comparison: 1% Colloidal Oatmeal Balm; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Paired t-test — The significance level threshold level was 0.05
Statistical Analysis 2: Comparison: EpiCeram Skin Barrier Emulsion; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Paired t-test — The significance level threshold level was 0.05
Statistical Analysis 3: Comparison: 1% Colloidal Oatmeal Balm vs EpiCeram Skin Barrier Emulsion; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.556, ANCOVA — The significance level threshold level was 0.05; Change from baseline as response, baseline score as covariate and treatment as factor; Mean Difference (Final Values) = -0.47, 95% CI 2-sided [-2.075 to 1.129], Standard Error of Mean 0.798

8. Primary Outcome: Change From Baseline in the Itch Assessment Score 7 Days After Treatment
Description: as for outcome 1
Time Frame: Baseline to seven days after treatment
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 40 | 12
units on a scale | 4.22 (2.815) | 6.53 (1.432)
Statistical Analysis 1: Comparison: 1% Colloidal Oatmeal Balm; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Paired t-test — The significance level threshold level was 0.05
Statistical Analysis 2: Comparison: EpiCeram Skin Barrier Emulsion; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Paired t-test — The significance level threshold level was 0.05
Statistical Analysis 3: Comparison: 1% Colloidal Oatmeal Balm vs EpiCeram Skin Barrier Emulsion; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.106, ANCOVA — The significance level threshold level was 0.05; Change from baseline as response, baseline score as covariate and treatment as factor; Mean Difference (Final Values) = -1.27, 95% CI 2-sided [-2.824 to 0.278], Standard Error of Mean 0.772

9. Secondary Outcome: Change From Baseline in Mean Corneometer Measurement Immediately Following Treatment
Description: Corneometer is a non-invasive instrument that measures hydration on the skin surface. During assessment, the corneometer was placed at a site adjacent to affected skin areas. Corneometer readings are directly related to the skin's electrical capacitance and increase as the skin becomes more hydrated.
Time Frame: Baseline to Immediately following treatment
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Mean (Standard Deviation); unit: arbitrary units
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 40 | 13
arbitrary units | 48.26 (24.913) | 21.71 (13.665)
Statistical Analysis 1: Comparison: 1% Colloidal Oatmeal Balm; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Paired t-test — The significance level threshold level was 0.05
Statistical Analysis 2: Comparison: EpiCeram Skin Barrier Emulsion; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Paired t-test — The significance level threshold level was 0.05
Statistical Analysis 3: Comparison: 1% Colloidal Oatmeal Balm vs EpiCeram Skin Barrier Emulsion; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANCOVA — The significance level threshold level was 0.05; Change from baseline as response, baseline score as covariate and treatment as factor; Mean Difference (Final Values) = 26.83, 95% CI 2-sided [13.407 to 40.247], Standard Error of Mean 6.681

10. Secondary Outcome: Change From Baseline in Mean Corneometer Measurement 1 Hour After Treatment
Description: as for outcome 9
Time Frame: Baseline to one hour after treatment
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Mean (Standard Deviation); unit: arbitrary units
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 40 | 13
arbitrary units | 27.00 (14.998) | 7.84 (7.881)
Statistical Analysis 1: Comparison: 1% Colloidal Oatmeal Balm; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Paired t-test — The significance level threshold level was 0.05
Statistical Analysis 2: Comparison: EpiCeram Skin Barrier Emulsion; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.004, Paired t-test — The significance level threshold level was 0.05
Statistical Analysis 3: Comparison: 1% Colloidal Oatmeal Balm vs EpiCeram Skin Barrier Emulsion; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANCOVA — The significance level threshold level was 0.05; Change from baseline as response, baseline score as covariate and treatment as factor; Mean Difference (Final Values) = 19.33, 95% CI 2-sided [11.301 to 27.352], Standard Error of Mean 3.996

11. Secondary Outcome: Change From Baseline in Mean Corneometer Measurement 2 Hours After Treatment
Description: as for outcome 9
Time Frame: Baseline to two hours after treatment
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Mean (Standard Deviation); unit: arbitrary units
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 40 | 13
arbitrary units | 23.20 (14.418) | 7.32 (8.525)
Statistical Analysis 1: Comparison: 1% Colloidal Oatmeal Balm; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Paired t-test — The significance level threshold level was 0.05
Statistical Analysis 2: Comparison: EpiCeram Skin Barrier Emulsion; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.009, Paired t-test — The significance level threshold level was 0.05
Statistical Analysis 3: Comparison: 1% Colloidal Oatmeal Balm vs EpiCeram Skin Barrier Emulsion; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANCOVA — The significance level threshold level was 0.05; Change from baseline as response, baseline score as covariate and treatment as factor; Mean Difference (Final Values) = 16.01, 95% CI 2-sided [7.829 to 24.187], Standard Error of Mean 4.072

12. Secondary Outcome: Change From Baseline in Mean Corneometer Measurement 3 Hours After Treatment
Description: as for outcome 9
Time Frame: Baseline to three hours after treatment
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Mean (Standard Deviation); unit: arbitrary units
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 38 | 13
arbitrary units | 21.05 (13.373) | 8.07 (7.706)
Statistical Analysis 1: Comparison: 1% Colloidal Oatmeal Balm; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Paired t-test — The significance level threshold level was 0.05
Statistical Analysis 2: Comparison: EpiCeram Skin Barrier Emulsion; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.003, Paired t-test — The significance level threshold level was 0.05
Statistical Analysis 3: Comparison: 1% Colloidal Oatmeal Balm vs EpiCeram Skin Barrier Emulsion; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANCOVA — The significance level threshold level was 0.05; Change from baseline as response, baseline score as covariate and treatment as factor; Mean Difference (Final Values) = 13.25, 95% CI 2-sided [5.684 to 20.820], Standard Error of Mean 3.764

13. Secondary Outcome: Change From Baseline in Mean Corneometer Measurement 4 Hours After Treatment
Description: as for outcome 9
Time Frame: Baseline to four hours after treatment
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Mean (Standard Deviation); unit: arbitrary units
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 40 | 13
arbitrary units | 19.65 (15.249) | 5.75 (9.491)
Statistical Analysis 1: Comparison: 1% Colloidal Oatmeal Balm; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Paired t-test — The significance level threshold level was 0.05
Statistical Analysis 2: Comparison: EpiCeram Skin Barrier Emulsion; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.049, Paired t-test — The significance level threshold level was 0.05
Statistical Analysis 3: Comparison: 1% Colloidal Oatmeal Balm vs EpiCeram Skin Barrier Emulsion; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.001, ANCOVA — The significance level threshold level was 0.05; Change from baseline as response, baseline score as covariate and treatment as factor; Mean Difference (Final Values) = 14.08, 95% CI 2-sided [5.766 to 22.387], Standard Error of Mean 4.138

14. Secondary Outcome: Change From Baseline in Mean Corneometer Measurement 5 Hours After Treatment
Description: as for outcome 9
Time Frame: Baseline to five hours after treatment
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Mean (Standard Deviation); unit: arbitrary units
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 40 | 13
arbitrary units | 21.48 (15.980) | 7.31 (10.205)
Statistical Analysis 1: Comparison: 1% Colloidal Oatmeal Balm; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Paired t-test — The significance level threshold level was 0.05
Statistical Analysis 2: Comparison: EpiCeram Skin Barrier Emulsion; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.024, Paired t-test — The significance level threshold level was 0.05
Statistical Analysis 3: Comparison: 1% Colloidal Oatmeal Balm vs EpiCeram Skin Barrier Emulsion; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.004, ANCOVA — The significance level threshold level was 0.05; Change from baseline as response, baseline score as covariate and treatment as factor; Mean Difference (Final Values) = 14.26, 95% CI 2-sided [4.862 to 23.660], Standard Error of Mean 4.679

15. Secondary Outcome: Change From Baseline in Mean Corneometer Measurement 6 Hours After Treatment
Description: as for outcome 9
Time Frame: Baseline to six hours after treatment
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Mean (Standard Deviation); unit: arbitrary units
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 40 | 13
arbitrary units | 18.71 (14.882) | 6.05 (7.687)
Statistical Analysis 1: Comparison: 1% Colloidal Oatmeal Balm; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Paired t-test — The significance level threshold level was 0.05
Statistical Analysis 2: Comparison: EpiCeram Skin Barrier Emulsion; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.015, Paired t-test — The significance level threshold level was 0.05
Statistical Analysis 3: Comparison: 1% Colloidal Oatmeal Balm vs EpiCeram Skin Barrier Emulsion; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.004, ANCOVA — The significance level threshold level was 0.05; Change from baseline as response, baseline score as covariate and treatment as factor; Mean Difference (Final Values) = 12.77, 95% CI 2-sided [4.291 to 21.252], Standard Error of Mean 4.222

16. Secondary Outcome: Change From Baseline in Mean Corneometer Measurement 7 Days After Treatment
Description: as for outcome 9
Time Frame: Baseline to seven days after treatment
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Mean (Standard Deviation); unit: arbitrary units
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 40 | 12
arbitrary units | 21.01 (19.743) | 7.99 (11.404)
Statistical Analysis 1: Comparison: 1% Colloidal Oatmeal Balm; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Paired t-test — The significance level threshold level was 0.05
Statistical Analysis 2: Comparison: EpiCeram Skin Barrier Emulsion; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.034, Paired t-test — The significance level threshold level was 0.05
Statistical Analysis 3: Comparison: 1% Colloidal Oatmeal Balm vs EpiCeram Skin Barrier Emulsion; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.037, ANCOVA — The significance level threshold level was 0.05; Change from baseline as response, baseline score as covariate and treatment as factor; Mean Difference (Final Values) = 12.71, 95% CI 2-sided [0.805 to 24.621], Standard Error of Mean 5.925

17. Secondary Outcome: Participant Questionnaire on Day 0 Pre-treatment - Distracted by Itchy Skin
Description: Questions were answered before treatment by the participant. The question is "I'm less distracted by my itchy skin"
Time Frame: 0 Days - Pre-treatment
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 40 | 13
percentage of participants
  Strongly agree | 7.5 | 0
  Somewhat agree | 7.5 | 0
  Neither agree or disagree | 7.5 | 0
  Somewhat disagree | 37.5 | 38.5
  Strongly disagree | 40.0 | 61.5
  I don't have an opinion | 0 | 0

18. Secondary Outcome: Participant Questionnaire on Day 0 Pre-treatment - Calmer Skin
Description: Questions were answered before treatment by the participant. The question is "I wake up to calmer skin"
Time Frame: 0 Days - Pre-treatment
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 40 | 13
percentage of participants
  Strongly agree | 10.0 | 7.7
  Somewhat agree | 10.0 | 23.1
  Neither agree or disagree | 5.0 | 0
  Somewhat disagree | 37.5 | 23.1
  Strongly disagree | 37.5 | 46.2
  I don't have an opinion | 0 | 0

19. Secondary Outcome: Participant Questionnaire on Day 0 Pre-treatment - Smooth Skin
Description: Questions were answered before treatment by the participant. The question is "My skin feels smooth"
Time Frame: 0 Days - Pre-treatment
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 40 | 13
percentage of participants
  Strongly agree | 2.5 | 0
  Somewhat agree | 2.5 | 0
  Neither agree or disagree | 10.0 | 7.7
  Somewhat disagree | 32.5 | 23.1
  Strongly disagree | 52.5 | 69.2
  I don't have an opinion | 0 | 0

20. Secondary Outcome: Participant Questionnaire on Day 0 Pre-treatment - Comfortable Showing Skin
Description: Questions were answered before treatment by the participant. The question is "I feel comfortable showing my skin"
Time Frame: 0 Days - Pre-treatment
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 40 | 13
percentage of participants
  Strongly agree | 15.0 | 0
  Somewhat agree | 5.0 | 7.7
  Neither agree or disagree | 12.5 | 30.8
  Somewhat disagree | 25.0 | 15.4
  Strongly disagree | 37.5 | 46.2
  I don't have an opinion | 5.0 | 0

21. Secondary Outcome: Participant Questionnaire on Day 0 Pre-treatment - Moisturized Skin
Description: Questions were answered before treatment by the participant. The question is "My skin feels moisturized"
Time Frame: 0 Days - Pre-treatment
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 40 | 13
percentage of participants
  Strongly agree | 0 | 0
  Somewhat agree | 5.0 | 0
  Neither agree or disagree | 7.5 | 0
  Somewhat disagree | 27.5 | 23.1
  Strongly disagree | 60.0 | 76.9
  I don't have an opinion | 0 | 0

22. Secondary Outcome: Participant Questionnaire on Day 0 Pre-treatment - Touchable Skin
Description: Questions were answered before treatment by the participant. The question is "My skin feels touchable"
Time Frame: 0 Days - Pre-treatment
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 40 | 13
percentage of participants
  Strongly agree | 7.5 | 7.7
  Somewhat agree | 10.0 | 7.7
  Neither agree or disagree | 7.5 | 7.7
  Somewhat disagree | 40.0 | 38.5
  Strongly disagree | 30.0 | 38.5
  I don't have an opinion | 5.0 | 0

23. Secondary Outcome: Participant Questionnaire on Day 0 Pre-treatment - Soft Skin
Description: Questions were answered before treatment by the participant. The question is "My skin feels soft"
Time Frame: 0 Days - Pre-treatment
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 40 | 13
percentage of participants
  Strongly agree | 2.5 | 0
  Somewhat agree | 2.5 | 7.7
  Neither agree or disagree | 10.0 | 15.4
  Somewhat disagree | 30.0 | 15.4
  Strongly disagree | 50.0 | 61.5
  I don't have an opinion | 5.0 | 0

24. Secondary Outcome: Participant Questionnaire on Day 0 Pre-treatment - Distracted by Itchy Eczema Skin Over Past 2 Days
Description: Questions were answered before treatment by the participant. The question is "Thinking about your experience over the past two days, please describe your degree of being distracted by your itchy, eczema skin. Would you say you were"
Time Frame: 0 Days - Pre-treatment
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 40 | 13
percentage of participants
  Not at all distracted | 2.5 | 0
  Slightly distracted | 7.5 | 0
  Moderately distracted | 35.0 | 23.1
  Very distracted | 37.5 | 61.5
  Extremely distracted | 17.5 | 15.4
  I don't have an opinion | 0 | 0

25. Secondary Outcome: Participant Questionnaire on Day 0 Pre-treatment - Skin Upon Waking Over Past 2 Days
Description: Questions were answered before treatment by the participant. The question is "Thinking about your experience over the past two days, how would you describe your skin upon awakening?"
Time Frame: 0 Days - Pre-treatment
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 40 | 13
percentage of participants
  Extremely calm | 2.5 | 7.7
  Very calm | 0 | 0
  Moderately calm | 22.5 | 15.4
  Slightly calm | 30.0 | 23.1
  Not at all calm | 35.0 | 53.8
  I don't have an opinion | 10.0 | 0

26. Secondary Outcome: Participant Questionnaire on Day 0 Pre-treatment - Sleep During Past 2 Days
Description: Questions were answered before treatment by the participant. The question is "Thinking about how well you slept during the past two days, would you say your sleep was?"
Time Frame: 0 Days - Pre-treatment
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 40 | 13
percentage of participants
  Very good | 5.0 | 0
  Moderately good | 25.0 | 23.1
  Neither bad nor good | 15.0 | 15.4
  Moderately bad | 37.5 | 46.2
  Very bad | 17.5 | 15.4
  I don't have an opinion | 0 | 0

27. Secondary Outcome: Participant Questionnaire on Day 0 Pre-treatment - Comfortable Showing Skin Over Past 2 Days
Description: Questions were answered before treatment by the participant. The question is "Thinking about how comfortable you felt showing your skin during the last two days, would you say that you were"
Time Frame: 0 Days - Pre-treatment
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 40 | 13
percentage of participants
  Extremely comfortable | 2.5 | 0
  Very comfortable | 2.5 | 0
  Moderately comfortable | 27.5 | 7.7
  Slightly comfortable | 30.0 | 23.1
  Not at all comfortable | 32.5 | 69.2
  I don't have an opinion | 5.0 | 0

28. Secondary Outcome: Participant Questionnaire Immediately After Treatment - Product Fast Absorbing
Description: Questions were answered immediately after treatment by the participant. The question is "This product is fast absorbing"
Time Frame: 0 Days - Immediately after treatment
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 40 | 13
percentage of participants
  Strongly agree | 22.5 | 53.8
  Somewhat agree | 42.5 | 38.5
  Neither agree or disagree | 15.0 | 0
  Somewhat disagree | 12.5 | 7.7
  Strongly disagree | 5.0 | 0
  I don't have an opinion | 2.5 | 0

29. Secondary Outcome: Participant Questionnaire Immediately After Treatment - Calm Skin
Description: Questions were answered immediately after treatment by the participant. The question is "This product calms my skin"
Time Frame: 0 Days - Immediately after treatment
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 40 | 13
percentage of participants
  Strongly agree | 30.0 | 53.8
  Somewhat agree | 37.5 | 38.5
  Neither agree or disagree | 15.0 | 7.7
  Somewhat disagree | 12.5 | 0
  Strongly disagree | 2.5 | 0
  I don't have an opinion | 2.5 | 0

30. Secondary Outcome: Participant Questionnaire Immediately After Treatment - Moisturized Skin
Description: Questions were answered immediately after treatment by the participant. The question is "This product leaves my skin feeling immediately moisturized"
Time Frame: 0 Days - Immediately after treatment
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 40 | 13
percentage of participants
  Strongly agree | 42.5 | 38.5
  Somewhat agree | 40.0 | 46.2
  Neither agree or disagree | 15.0 | 7.7
  Somewhat disagree | 2.5 | 7.7
  Strongly disagree | 0 | 0
  I don't have an opinion | 0 | 0

31. Secondary Outcome: Participant Questionnaire Immediately After Treatment - Product Does Not Sting
Description: Questions were answered immediately after treatment by the participant. The question is "This product does not sting when applied"
Time Frame: 0 Days - Immediately after treatment
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 40 | 13
percentage of participants
  Strongly agree | 50.0 | 53.8
  Somewhat agree | 32.5 | 7.7
  Neither agree or disagree | 2.5 | 0
  Somewhat disagree | 10.0 | 23.1
  Strongly disagree | 5.0 | 15.4
  I don't have an opinion | 0 | 0

32. Secondary Outcome: Participant Questionnaire 4 Hours After Treatment - Long Lasting Moisture
Description: Questions were answered four hours after treatment by the participant. The question is "This product provides long lasting moisture"
Time Frame: Four hours after treatment
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 40 | 13
percentage of participants
  Strongly agree | 55.0 | 38.5
  Somewhat agree | 25.0 | 46.2
  Neither agree or disagree | 2.5 | 0
  Somewhat disagree | 10.0 | 7.7
  Strongly disagree | 5.0 | 7.7
  I don't have an opinion | 2.5 | 0

33. Secondary Outcome: Participant Questionnaire 4 Hours After Treatment - Skin Feeling Soft
Description: Questions were answered four hours after treatment by the participant. The question is "This product leaves my skin feeling soft"
Time Frame: Four hours after treatment
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 40 | 13
percentage of participants
  Strongly agree | 40.0 | 46.2
  Somewhat agree | 45.0 | 38.5
  Neither agree or disagree | 7.5 | 0
  Somewhat disagree | 5.0 | 0
  Strongly disagree | 0 | 15.4
  I don't have an opinion | 2.5 | 0

34. Secondary Outcome: Participant Questionnaire 5 Hours After Treatment - Long Lasting Moisture
Description: Questions were answered five hours after treatment by the participant. The question is "This product provides long lasting moisture"
Time Frame: Five hours after treatment
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 40 | 13
percentage of participants
  Strongly agree | 60.0 | 61.5
  Somewhat agree | 27.5 | 30.8
  Neither agree or disagree | 2.5 | 0
  Somewhat disagree | 2.5 | 7.7
  Strongly disagree | 5.0 | 0
  I don't have an opinion | 2.5 | 0

35. Secondary Outcome: Participant Questionnaire 5 Hours After Treatment - Skin Feeling Soft
Description: Questions were answered five hours after treatment by the participant. The question is "This product leaves my skin feeling soft"
Time Frame: Five hours after treatment
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 40 | 13
percentage of participants
  Strongly agree | 47.5 | 53.8
  Somewhat agree | 35.0 | 30.8
  Neither agree or disagree | 2.5 | 7.7
  Somewhat disagree | 7.5 | 7.7
  Strongly disagree | 2.5 | 0
  I don't have an opinion | 5.0 | 0

36. Secondary Outcome: Participant Questionnaire 6 Hours After Treatment - Long Lasting Moisture
Description: Questions were answered six hours after treatment by the participant. The question is "This product provides long lasting moisture"
Time Frame: Six hours after treatment
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 40 | 13
percentage of participants
  Strongly agree | 60.0 | 38.5
  Somewhat agree | 27.5 | 53.8
  Neither agree or disagree | 2.5 | 0
  Somewhat disagree | 10.0 | 0
  Strongly disagree | 0 | 7.7
  I don't have an opinion | 0 | 0

37. Secondary Outcome: Participant Questionnaire 6 Hours After Treatment - Calms Skin
Description: Questions were answered six hours after treatment by the participant. The question is "This product calms my skin"
Time Frame: Six hours after treatment
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 40 | 13
percentage of participants
  Strongly agree | 47.5 | 61.5
  Somewhat agree | 35.0 | 30.8
  Neither agree or disagree | 7.5 | 7.7
  Somewhat disagree | 7.5 | 0
  Strongly disagree | 2.5 | 0
  I don't have an opinion | 0 | 0

38. Secondary Outcome: Participant Questionnaire 6 Hours After Treatment - Distracted by Itchy Skin
Description: Questions were answered six hours after treatment by the participant. The question is "I'm less distracted by my itchy skin"
Time Frame: Six hours after treatment
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 40 | 13
percentage of participants
  Strongly agree | 52.5 | 53.8
  Somewhat agree | 27.5 | 38.5
  Neither agree or disagree | 12.5 | 7.7
  Somewhat disagree | 7.5 | 0
  Strongly disagree | 0 | 0
  I don't have an opinion | 0 | 0

39. Secondary Outcome: Participant Questionnaire 6 Hours After Treatment - Comfortable Showing Skin
Description: Questions were answered six hours after treatment by the participant. The question is "I feel comfortable showing my skin"
Time Frame: Six hours after treatment
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 40 | 13
percentage of participants
  Strongly agree | 35.0 | 38.5
  Somewhat agree | 30.0 | 38.5
  Neither agree or disagree | 15.0 | 7.7
  Somewhat disagree | 12.5 | 7.7
  Strongly disagree | 5.0 | 7.7
  I don't have an opinion | 2.5 | 0

40. Secondary Outcome: Participant Questionnaire 6 Hours After Treatment - Shield for Skin
Description: Questions were answered six hours after treatment by the participant. The question is "This product feels like a shield for my skin"
Time Frame: Six hours after treatment
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 40 | 13
percentage of participants
  Strongly agree | 37.5 | 38.5
  Somewhat agree | 37.5 | 61.5
  Neither agree or disagree | 17.5 | 0
  Somewhat disagree | 7.5 | 0
  Strongly disagree | 0 | 0
  I don't have an opinion | 0 | 0

41. Secondary Outcome: Participant Questionnaire 6 Hours After Treatment - Skin Feels Moisturized
Description: Questions were answered six hours after treatment by the participant. The question is "This product leaves my skin feeling moisturized"
Time Frame: Six hours after treatment
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 40 | 13
percentage of participants
  Strongly agree | 57.5 | 46.2
  Somewhat agree | 27.5 | 38.5
  Neither agree or disagree | 2.5 | 7.7
  Somewhat disagree | 10.0 | 7.7
  Strongly disagree | 0 | 0
  I don't have an opinion | 2.5 | 0

42. Secondary Outcome: Participant Questionnaire 6 Hours After Treatment - Skin Feels Touchable
Description: Questions were answered six hours after treatment by the participant. The question is "This product makes my skin feel touchable"
Time Frame: Six hours after treatment
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 40 | 13
percentage of participants
  Strongly agree | 42.5 | 61.5
  Somewhat agree | 35.0 | 15.4
  Neither agree or disagree | 5.0 | 7.7
  Somewhat disagree | 12.5 | 15.4
  Strongly disagree | 2.5 | 0
  I don't have an opinion | 2.5 | 0

43. Secondary Outcome: Participant Questionnaire 6 Hours After Treatment - Skin Feels Soft
Description: Questions were answered six hours after treatment by the participant. The question is "This product makes my skin feel soft"
Time Frame: Six hours after treatment
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 40 | 13
percentage of participants
  Strongly agree | 50.0 | 53.8
  Somewhat agree | 30.0 | 30.8
  Neither agree or disagree | 10.0 | 0
  Somewhat disagree | 5.0 | 7.7
  Strongly disagree | 2.5 | 7.7
  I don't have an opinion | 2.5 | 0

44. Secondary Outcome: Participant Questionnaire 6 Hours After Treatment - Skin Feels Smooth
Description: Questions were answered six hours after treatment by the participant. The question is "This product leaves my skin feeling smooth"
Time Frame: Six hours after treatment
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 40 | 13
percentage of participants
  Strongly agree | 45.0 | 53.8
  Somewhat agree | 32.5 | 30.8
  Neither agree or disagree | 7.5 | 0
  Somewhat disagree | 5.0 | 7.7
  Strongly disagree | 7.5 | 7.7
  I don't have an opinion | 2.5 | 0

45. Secondary Outcome: Participant Questionnaire 6 Hours After Treatment - Degree of Distraction by Itchy Eczema Skin
Description: Questions were answered six hours after treatment by the participant. The question is "Thinking about your experience after using this product, please describe your degree of being distracted by your itchy, eczema skin. Would you say you were"
Time Frame: Six hours after treatment
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 40 | 13
percentage of participants
  Not at all distracted | 35.0 | 23.1
  Slightly distracted | 40.0 | 46.2
  Moderately distracted | 17.5 | 15.4
  Very distracted | 7.5 | 15.4
  Extremely distracted | 0 | 0
  I don't have an opinion | 0 | 0

46. Secondary Outcome: Participant Questionnaire 6 Hours After Treatment - Degree of Comfortableness Showing Skin
Description: Questions were answered six hours after treatment by the participant. The question is "Thinking about how comfortable you felt showing your skin after using this product, would you say that you were"
Time Frame: Six hours after treatment
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 40 | 13
percentage of participants
  Extremely comfortable | 22.5 | 23.1
  Very comfortable | 27.5 | 30.8
  Moderately comfortable | 40.0 | 30.8
  Slightly comfortable | 2.5 | 7.7
  Not at all comfortable | 2.5 | 7.7
  I don't have an opinion | 5.0 | 0

47. Secondary Outcome: Participant Questionnaire 7 Days After Treatment - Skin Feels Calm
Description: Questions were answered seven days after treatment by the participant. The question is "This product calms my skin"
Time Frame: Seven days after treatment
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 40 | 12
percentage of participants
  Strongly agree | 60.0 | 66.7
  Somewhat agree | 32.5 | 33.3
  Neither agree or disagree | 0 | 0
  Somewhat disagree | 2.5 | 0
  Strongly disagree | 5.0 | 0
  I don't have an opinion | 0 | 0

48. Secondary Outcome: Participant Questionnaire 7 Days After Treatment - Distracted by Itchy Skin
Description: Questions were answered seven days after treatment by the participant. The question is "I'm less distracted by my itchy skin"
Time Frame: Seven days after treatment
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 40 | 12
percentage of participants
  Strongly agree | 55.0 | 83.3
  Somewhat agree | 32.5 | 16.7
  Neither agree or disagree | 2.5 | 0
  Somewhat disagree | 2.5 | 0
  Strongly disagree | 7.5 | 0
  I don't have an opinion | 0 | 0

49. Secondary Outcome: Participant Questionnaire 7 Days After Treatment - Calmer Skin on Waking
Description: Questions were answered seven days after treatment by the participant. The question is "I wake up to calmer skin"
Time Frame: Seven days after treatment
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 40 | 12
percentage of participants
  Strongly agree | 65.0 | 66.7
  Somewhat agree | 20.0 | 25.0
  Neither agree or disagree | 5.0 | 0
  Somewhat disagree | 2.5 | 0
  Strongly disagree | 7.5 | 8.3
  I don't have an opinion | 0 | 0

50. Secondary Outcome: Participant Questionnaire 7 Days After Treatment - Comfortable Showing Skin
Description: Questions were answered seven days after treatment by the participant. The question is "I feel comfortable showing my skin"
Time Frame: Seven days after treatment
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 40 | 12
percentage of participants
  Strongly agree | 42.5 | 50.0
  Somewhat agree | 32.5 | 41.7
  Neither agree or disagree | 7.5 | 0
  Somewhat disagree | 12.5 | 8.3
  Strongly disagree | 5.0 | 0
  I don't have an opinion | 0 | 0

51. Secondary Outcome: Participant Questionnaire 7 Days After Treatment - Long Lasting Moisture
Description: Questions were answered seven days after treatment by the participant. The question is "This product provides long lasting moisture to my skin"
Time Frame: Seven days after treatment
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 40 | 12
percentage of participants
  Strongly agree | 65.0 | 50.0
  Somewhat agree | 22.5 | 41.7
  Neither agree or disagree | 2.5 | 0
  Somewhat disagree | 2.5 | 8.3
  Strongly disagree | 7.5 | 0
  I don't have an opinion | 0 | 0

52. Secondary Outcome: Participant Questionnaire 7 Days After Treatment - Shield for Skin
Description: Questions were answered seven days after treatment by the participant. The question is "This product feels like a shield for my skin"
Time Frame: Seven days after treatment
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 40 | 12
percentage of participants
  Strongly agree | 52.5 | 66.7
  Somewhat agree | 30.0 | 25.0
  Neither agree or disagree | 12.5 | 8.3
  Somewhat disagree | 0 | 0
  Strongly disagree | 2.5 | 0
  I don't have an opinion | 2.5 | 0

53. Secondary Outcome: Participant Questionnaire 7 Days After Treatment - Skin Feels Moisturized
Description: Questions were answered seven days after treatment by the participant. The question is "This product leaves my skin feeling moisturized"
Time Frame: Seven days after treatment
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 40 | 12
percentage of participants
  Strongly agree | 72.5 | 50.0
  Somewhat agree | 22.5 | 50.0
  Neither agree or disagree | 0 | 0
  Somewhat disagree | 0 | 0
  Strongly disagree | 5.0 | 0
  I don't have an opinion | 0 | 0

54. Secondary Outcome: Participant Questionnaire 7 Days After Treatment - Skin Feels Touchable
Description: Questions were answered seven days after treatment by the participant. The question is "This product makes my skin feel touchable"
Time Frame: Seven days after treatment
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 40 | 12
percentage of participants
  Strongly agree | 57.5 | 41.7
  Somewhat agree | 22.5 | 58.3
  Neither agree or disagree | 5.0 | 0
  Somewhat disagree | 10.0 | 0
  Strongly disagree | 5.0 | 0
  I don't have an opinion | 0 | 0

55. Secondary Outcome: Participant Questionnaire 7 Days After Treatment - Product Does Not Rub Off on Sheets
Description: Questions were answered seven days after treatment by the participant. The question is "This product does not rub off on sheets"
Time Frame: Seven days after treatment
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 40 | 12
percentage of participants
  Strongly agree | 42.5 | 83.3
  Somewhat agree | 25.0 | 16.7
  Neither agree or disagree | 10.0 | 0
  Somewhat disagree | 10.0 | 0
  Strongly disagree | 12.5 | 0
  I don't have an opinion | 0 | 0

56. Secondary Outcome: Participant Questionnaire 7 Days After Treatment - Skin Feels Soft
Description: Questions were answered seven days after treatment by the participant. The question is "This product makes my skin feel soft"
Time Frame: Seven days after treatment
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 40 | 12
percentage of participants
  Strongly agree | 65.0 | 50.0
  Somewhat agree | 27.5 | 50.0
  Neither agree or disagree | 2.5 | 0
  Somewhat disagree | 0 | 0
  Strongly disagree | 5.0 | 0
  I don't have an opinion | 0 | 0

57. Secondary Outcome: Participant Questionnaire 7 Days After Treatment - Moisturized All Day
Description: Questions were answered seven days after treatment by the participant. The question is "This product leaves my skin feeling moisturized all day"
Time Frame: Seven days after treatment
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 40 | 12
percentage of participants
  Strongly agree | 67.5 | 33.3
  Somewhat agree | 17.5 | 50.0
  Neither agree or disagree | 2.5 | 0
  Somewhat disagree | 7.5 | 16.7
  Strongly disagree | 5.0 | 0
  I don't have an opinion | 0 | 0

58. Secondary Outcome: Participant Questionnaire 7 Days After Treatment - Slept Better
Description: Questions were answered seven days after treatment by the participant. The question is "I slept better due to less itching or skin discomfort"
Time Frame: Seven days after treatment
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 40 | 12
percentage of participants
  Strongly agree | 45.0 | 41.7
  Somewhat agree | 30.0 | 58.3
  Neither agree or disagree | 17.5 | 0
  Somewhat disagree | 5.0 | 0
  Strongly disagree | 2.5 | 0
  I don't have an opinion | 0 | 0

59. Secondary Outcome: Participant Questionnaire 7 Days After Treatment - Skin Feels Smooth
Description: Questions were answered seven days after treatment by the participant. The question is "This product leaves my skin feeling smooth"
Time Frame: Seven days after treatment
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 40 | 12
percentage of participants
  Strongly agree | 60.0 | 66.7
  Somewhat agree | 27.5 | 25.0
  Neither agree or disagree | 2.5 | 0
  Somewhat disagree | 5.0 | 8.3
  Strongly disagree | 5.0 | 0
  I don't have an opinion | 0 | 0

60. Secondary Outcome: Participant Questionnaire 7 Days After Treatment - Degree of Distraction by Itchy Eczema Skin
Description: Questions were answered seven days after treatment by the participant. The question is "Thinking about your experience while using this product, please describe your degree of being distracted by your itchy, eczema skin. Would you say you were"
Time Frame: Seven days after treatment
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 39 | 12
percentage of participants
  Not at all distracted | 33.3 | 33.3
  Slightly distracted | 56.4 | 50.0
  Moderately distracted | 5.1 | 0
  Very distracted | 0 | 0
  Extremely distracted | 5.1 | 16.7
  I don't have an opinion | 0 | 0

61. Secondary Outcome: Participant Questionnaire 7 Days After Treatment - Skin on Waking
Description: Questions were answered seven days after treatment by the participant. The question is "Thinking about your experience when using this product, how would you describe your skin upon awakening?"
Time Frame: Seven days after treatment
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 40 | 12
percentage of participants
  Extremely calm | 32.5 | 8.3
  Very calm | 30.0 | 58.3
  Moderately calm | 27.5 | 25.0
  Slightly calm | 5.0 | 0
  Not at all calm | 5.0 | 8.3
  I don't have an opinion | 0 | 0

62. Secondary Outcome: Participant Questionnaire 7 Days After Treatment - Degree of Sleep
Description: Questions were answered seven days after treatment by the participant. The question is "Thinking about how well you slept when using this product, would you say your sleep was?"
Time Frame: 7 days after treatment
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 40 | 12
percentage of participants
  Very good | 45.0 | 50.0
  Moderately good | 30.0 | 50.0
  Neither bad nor good | 20.0 | 0
  Moderately bad | 2.5 | 0
  Very bad | 2.5 | 0
  I don't have an opinion | 0 | 0

63. Secondary Outcome: Participant Questionnaire 7 Days After Treatment - Degree of Comfortableness Showing Skin
Description: Questions were answered seven days after treatment by the participant. The question is "Thinking about how comfortable you felt showing your skin while using this product, would you say that you were"
Time Frame: Seven days after treatment
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 40 | 12
percentage of participants
  Extremely comfortable | 25.0 | 25.0
  Very comfortable | 37.5 | 33.3
  Moderately comfortable | 17.5 | 33.3
  Slightly comfortable | 17.5 | 8.3
  Not at all comfortable | 2.5 | 0
  I don't have an opinion | 0 | 0

ADVERSE EVENTS:
Time Frame: Day 7 ± 1 day, +30 days for serious adverse events.
Description: Adverse events were systematically collected beginning with the signing of the informed consent form and continuing at each study visit through Visit 3 (Day 7 ± 1 day). Serious adverse events were reported through 30 days after product use. Spontaneously reported adverse events collected outside of the regularly scheduled visits were also recorded.
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/13
Other Adverse Events (participants affected / at risk) | 6/40 | 1/13
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 1% Colloidal Oatmeal Balm (N=40) | EpiCeram Skin Barrier Emulsion (N=13)
Application Site Pain (General disorders) | 6 | 0
Pain (General disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal investigators agreed not to publish the study results without prior sponsor approval.